CLINICAL TRIAL: NCT03725449
Title: An Online Intervention for Skin Self-Checks Among Individuals at Increased Risk for Melanoma
Brief Title: Internet-based Intervention for Skin Self-Examination in Participants With Increased Risk for Melanoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sharon Manne, PhD, Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro20170000597; NCI-2018-02006 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Pro20170000597; 131707 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH)
Record Dates: First submitted 2018-10-01; First posted 2018-10-31 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Dysplastic Nevus; Health Status Unknown; Melanoma; No Evidence of Disease
MeSH Terms: conditions — Dysplastic Nevus Syndrome; Melanoma | interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase I (user testing) (Experimental): Participants complete telephone-based usability testing of the online program. Participants complete between 1-5 user testing sessions of the mySmartCheck program (about 45-60 minutes per session) to provide feedback on acceptability, satisfaction, comprehension, and usability.
  Interventions: Behavioral: mySmartCheck
- Phase II Group I (mySmartCheck) (Experimental): Participants are asked to complete a baseline survey. After completing the baseline survey, participants receive access to mySmartCheck program, and continue to receive standard of care. Participants are asked to complete another survey 13 weeks post-baseline.
  Interventions: Other: Best Practice; Other: Survey Administration
- Phase II Group II (standard of care) (Experimental): Participants are asked to complete a baseline survey. After completing the baseline survey, participants receive standard of care. Participants are asked to complete another survey 13 weeks post-baseline.
  Interventions: Other: Best Practice; Other: Survey Administration

INTERVENTIONS:
Other: Best Practice — Receive standard of care
  Other Names: standard of care; standard therapy
  Arms: Phase II Group I (mySmartCheck); Phase II Group II (standard of care)
Behavioral: mySmartCheck — Receive access to mySmartcheck program
  Arms: Phase I (user testing)
Other: Survey Administration — Ancillary studies
  Arms: Phase II Group I (mySmartCheck); Phase II Group II (standard of care)

SUMMARY:
This trial studies an internet-based intervention for skin self-examination (SSE) in participants at increased risk for melanoma. Early detection of suspicious growths on the skin can be done by performing regular SSE checks. Using an internet-based intervention, such as mySmartCheck, may help to promote regular, thorough checks on the skin in individuals at increased risk for melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the impact of mySmartCheck versus usual care on skin-self-examination (SSE) behaviors among individuals at increased risk for developing melanoma.

SECONDARY OBJECTIVES:

I. To evaluate the impact of mySmartCheck versus usual care on patients barriers and benefits to conducting SSE, SSE self-efficacy (confidence), level of worry about developing melanoma, and number of health care consultations (visits, telephone calls, and emails).

II. To evaluate whether mySmartCheck effects are moderated by the patient's Total Body Photography (TBP) status.

III. To identify barriers and facilitators to using mySmartCheck.

OUTLINE:

PHASE I: Participants complete a telephone based usability testing of the online program. Participants complete between 1-5 user testing sessions of the mySmartCheck program (about 45-60 minutes per session) to provide feedback on acceptability, satisfaction, comprehension, and usability.

PHASE II: Participants are randomized to 1 of 2 groups. Both the intervention and control group complete a baseline survey as well as a 13 weeks post-baseline survey.

GROUP I: After completing the baseline survey, participants receive access to the mySmartCheck program, and continue to receive standard of care. Participants are asked to complete another survey 13 weeks post-baseline.

GROUP II: After completing the baseline survey, participants receive standard of care. Participants are asked to complete another survey 13 weeks post-baseline.

Study duration is 13 weeks for all participants.

ELIGIBILITY:
Inclusion Criteria:

* At increased risk for melanoma due to a personal history of treated melanoma without current evidence of disease, a family history of melanoma in a first-degree relative, and/or having a high-risk mole phenotype (i.e., >= 50 normal moles or >= 1 abnormal mole [dysplastic nevus]).
* Access to a computer connected to the Internet.
* Not adherent to SSE recommendations (i.e., did not conduct a thorough SSE during each of the previous 3 months).
* Able to speak and read English.
* Able to provide informed consent.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2018-11-03 (Actual); Primary Completion 2020-08-29 (Actual); Study Completion 2020-08-29 (Actual)

PRIMARY OUTCOMES:
Performance of thorough skin-self examination (SSE) | Up to 13 weeks
  Thorough SSE is defined as thoroughly examining each area of the body during the most recent SSE skin self-check in the past 2 months

SECONDARY OUTCOMES:
Performance of thorough SSE in the past 1 month | Up to 13 weeks
  Thorough SSE is defined as thoroughly examining each area of the body during the most recent SSE skin self-check in the past 1 month
Number of SSEs performed (regardless of thoroughness) | Up to 13 weeks
  The total number of self-reported SSEs performed (regardless of their thoroughness)
Number of body areas examined during SSE | Up to 13 weeks
  The number of body areas (out of 15 total) examined during each SSE will be recorded.
Benefits to SSE | Up to 13 weeks
  The impact of mySmartCheck on patients' benefits to conducting SSE will be examined using 7 items.
Barriers to SSE | Up to 13 weeks
  The impact of mySmartCheck on patients' barriers to conducting SSE will be examined using 10 items.
SSE self-efficacy | Up to 13 weeks
  The impact of MySmartCheck on patient's SSE self-efficacy will be examined using 9 items.
Level of worry about melanoma | Up to 13 weeks
  The impact of mySmartCheck on patients' level of worry about melanoma will be examined using 2 items.
Number of health care consultations | Up to 13 weeks
  Survey questions will ask about the number of health care consultations related to skin cancer surveillance in the past 3 months. Questions will include consultation reasons and outcomes.
Barriers and facilitators to using mySmart check | Up to 13 weeks
  Three multi-item scales will be used to measure barriers and facilitators to using the mySmartCheck program. The first scale is 15 items (5-point response scale from "not at all" to "a lot") adapted from The Internet Impact and Effectiveness Questionnaire. This scale measures patients' perceptions of an Internet intervention in terms of the program's effectiveness in resolving their targeted health condition. The second scale includes 18 items (3-point response scale from "not a problem" to "a major problem") adapted from the Internet Intervention Adherence Questionnaire. This scale is used to identify obstacles and barriers that interfere with using Internet intervention programs. The final scale includes 13 items (4-point response scale from "not at all" to "very") adapted from the Internet Evaluation and Utility Questionnaire. This scale measures patients' experiences and perceptions of an Internet intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Manne, PhD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States

REFERENCES:
- [Derived] Manne SL, Marchetti MA, Kashy DA, Heckman CJ, Ritterband LM, Thorndike FP, Viola A, Lozada C, Coups EJ. mySmartCheck, a Digital Intervention to Promote Skin Self-examination Among Individuals Diagnosed With or at Risk for Melanoma: A Randomized Clinical Trial. Ann Behav Med. 2022 Aug 2;56(8):791-803. doi: 10.1093/abm/kaab090. PMID 34637495